CLINICAL TRIAL: NCT02071420
Title: Efficacy of a Combined Ergonomic Health Promotion Intervention on Employee Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Lucas Carr, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201306711
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Sedentary; Overweight
MeSH Terms: conditions — Sedentary Behavior; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): This group will receive the seated active workstation intervention, the ergonomic intervention and the email intervention for 16 weeks.
  Interventions: Behavioral: Active Workstation Intervention; Behavioral: Ergonomic Intervention; Behavioral: Email Intervention; Device: Bluetooth enabled device (Wahoo Fitness Blue SC sensor) and accompanying iPod application.
- Active Control (Active Comparator): This group will receive the ergonomic intervention and email intervention only for 16 weeks. This group will not receive a seated active workstation.
  Interventions: Behavioral: Ergonomic Intervention; Behavioral: Email Intervention; Device: Bluetooth enabled device (Wahoo Fitness Blue SC sensor) and accompanying iPod application.

INTERVENTIONS:
Behavioral: Active Workstation Intervention — Participants in the experimental group will receive a seated active workstation at their work setting for 16 weeks.
  Arms: Experimental Group
Behavioral: Ergonomic Intervention — Participants of both arms will receive a face to face ergonomic workstation optimization intervention. This consultation will take 30 minutes to complete and will be performed at the participant's actual work station.
Behavioral: Email Intervention — Participants of both arms will receive three emails per week for 16 weeks. Messages will be consistent with what they hear in the ergonomic intervention (e.g., encourage taking breaks from sitting at work and adjusting posture to be in line with ergonomic principles).
Device: Bluetooth enabled device (Wahoo Fitness Blue SC sensor) and accompanying iPod application.

SUMMARY:
Our objective in this pilot study is to test the combined effect of a) replacing office workers' sedentary workstations with active workstations (LifeBalance Station) and b) optimizing computer workstation ergonomics on daily occupational sedentary time, cardiometabolic risk factors, musculoskeletal symptom health outcomes and work productivity.

DETAILED DESCRIPTION:
Primary Aim: To compare the effects of providing sedentary employees with seated active workstations in combination with an ergonomic intervention and regular motivational emails (experimental group) against the ergonomic intervention and regular emails only (active control group) on occupational sedentary behavior over 16 weeks.

Hypothesis: The addition of a seated active workstation will result in significant reductions in daily occupational sedentary time compared to the active control group.

Secondary Aims: To compare the effects of the experimental group against the active control group on secondary measures of cardiometabolic disease risk factors, musculoskeletal discomfort, cognitive function and work productivity.

Hypothesis 1: The experimental group will result in reduced cardiometabolic disease risk, musculoskeletal discomfort and work limitations compared to the active control group.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit overweight/obese (body mass index 25.0-40.0 kg/m2) adults (18-65 years) working in full-time (minimum 35 hours/week), sedentary (self-report sitting >75% work time) occupations at an independent work site.

Exclusion Criteria:

* Working in an office that will not meet the space or electrical requirements of the active workstation, acute or chronic illness not under treatment of a provider, orthopedic limitations that prohibit physical activity, current or planned pregnancy, hospitalization from a physical or mental disorder in the past six months and/or taking medication that may impair physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Carr, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Carr LJ, Leonhard C, Tucker S, Fethke N, Benzo R, Gerr F. Total Worker Health Intervention Increases Activity of Sedentary Workers. Am J Prev Med. 2016 Jan;50(1):9-17. doi: 10.1016/j.amepre.2015.06.022. Epub 2015 Aug 7. PMID 26260492

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: This group will receive the seated active workstation intervention, the ergonomic intervention and the email intervention for 16 weeks.
  Active Workstation Intervention: Participants in the experimental group will receive a seated active workstation at their work setting for 16 weeks.
  Ergonomic Intervention: Participants of both arms will receive a face to face ergonomic workstation optimization intervention. This consultation will take 30 minutes to complete and will be performed at the participant's actual work station.
  Email Intervention: Participants of both arms will receive three emails per week for 16 weeks. Messages will be consistent with what they hear in the ergonomic intervention (e.g., encourage taking breaks from sitting at work and adjusting posture to be in line with ergonomic principles).
  Bluetooth enabled device (Wahoo Fitness Blue SC sensor) and accompanying iPod application.
- Active Control: This group will receive the ergonomic intervention and email intervention only for 16 weeks. This group will not receive a seated active workstation.
  Ergonomic Intervention: Participants of both arms will receive a face to face ergonomic workstation optimization intervention. This consultation will take 30 minutes to complete and will be performed at the participant's actual work station.
  Email Intervention: Participants of both arms will receive three emails per week for 16 weeks. Messages will be consistent with what they hear in the ergonomic intervention (e.g., encourage taking breaks from sitting at work and adjusting posture to be in line with ergonomic principles).
  Bluetooth enabled device (Wahoo Fitness Blue SC sensor) and accompanying iPod application.
Period: Overall Study
Arm/Group | Experimental Group | Active Control
Started | 30 | 30
Completed | 27 | 27
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Active Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (10.9) | 45.0 (10.7) | 45.1 (10.8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 21 | 21 | 42
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Occupational Physical Activity From Baseline to 16 Weeks
Description: Occupational physical activity (primary outcome) will be measured objectively with the GENEActiv physical activity monitor. The monitor will be worn on the right ankle and will be worn for 5 working days during all non-bathing hours. The outcome measure will be change in occupational activity (average counts/work day) from baseline to 16 weeks. The measure will be calculated as follows: 16 weeks value - baseline value.
Time Frame: Baseline and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Average counts/work day
Arm/Group | Experimental Group | Active Control
Number analyzed (Participants) | 27 | 27
Average counts/work day | 9752 [1067 to 18463] | -142 [-10623 to 10339]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 16 weeks during the intervention.
Arm/Group | Experimental Group | Active Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No